CLINICAL TRIAL: NCT00916136
Title: Evaluation of Skeletal Versus Cutaneous Traction for Diaphyseal Femur Fractures
Brief Title: Skeletal Versus Cutaneous Traction For Treatment of Femur Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 081299
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Femur Fracture
Keywords: Pre-operative Traction; Traction; Proximal Femur Fracture; Femoral Fractures; Femoral Fracture; Skeletal Traction; Cutaneous Traction
MeSH Terms: conditions — Femoral Fractures; Proximal Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cutaneous Traction (Active Comparator): Applied by using a strap on boot that attaches to the leg. A rope is attached to the boot. Weight is attached to the rope to use gravity to pull traction. The traction is left in place until patient is taken to surgery for reduction of the femur fracture.
  Interventions: Procedure: Femoral Traction
- Skeletal Traction (Active Comparator): A small incision is made on the inside of the knee and a pin is surgically inserted through the bone. Weights are then attached that will pull traction on the broken femur. This traction pin will stay in until patient is taken to surgery for reduction of the femur fracture.
  Interventions: Procedure: Femoral Traction

INTERVENTIONS:
Procedure: Femoral Traction — Femoral Traction is a temporary intervention to realign the broken bone and help relieve pressure and muscle spasms until operative fixation.
  Other Names: Bucks Traction; Traction Pins; Cutaneous Traction; Skeletal Traction; Skin Traction; Balance Skeletal Traction; Balanced Suspension Traction; (BST); Bryant's Traction; 90-degree Traction

SUMMARY:
The purpose of this study is to determine whether there are any differences in skeletal or cutaneous traction for the treatment of femur fractures.

DETAILED DESCRIPTION:
Diaphyseal femur fractures are a common occurrence in busy level one trauma centers and even in the age of damage control orthopaedics most of these fractures are fixed definitively within 24 hours. The historical method of temporizing these fractures has been to place a distal femoral or proximal tibial skeletal traction pin. However, in the pediatric population skeletal traction is not utilized due to concern for physeal injury and cutaneous traction has been the gold standard for decades. Reasons for skeletal traction in adults are not well defined and there are no clinical studies showing that skeletal traction provides better outcomes in time of reduction in the operating theater or better pain control than cutaneous traction. With the ever increasing amount of high energy trauma seen by junior residents in the emergency department time constraints have become a large factor in patient care. Long delays for sedation and equipment procurement make stabilizing a diaphyseal femur fracture a time consuming experience. The purpose of this study is to determine whether differences exist between skeletal and cutaneous femoral traction in terms of: 1) time in patient consultation and fracture stabilization; 2) cost and risk to the patient due to lack of conscious sedation; 3) pain scores prior to surgery; 4) time of reduction of the diaphyseal femur fraction during surgical fixation; and 5) pain relief after traction application.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to consent
* 18 years of age or older
* Sustained a diaphyseal femur fracture, open or closed
* English competent
* Isolated fracture on that extremity

Exclusion Criteria:

* Pathologic fracture
* Sedated patient
* Polytrauma to same extremity
* Unable or not willing to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Even, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Parker MJ, Handoll HH. Pre-operative traction for fractures of the proximal femur in adults. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD000168. doi: 10.1002/14651858.CD000168.pub2. PMID 16855952

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cutaneous Traction | Skeletal Traction
Started | 37 | 29
Completed | 37 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cutaneous Traction | Skeletal Traction | Total
Number analyzed (Participants) | 37 | 29 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 29 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (12.75) | 28.0 (13.5) | 27 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 30 | 24 | 54
Region of Enrollment [Number; unit: participants]
  United States | 37 | 29 | 66

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Two Groups in Regards to Resident Time.
Description: Time from consult entered to time traction apparatus is applied.
Time Frame: while in Emergency Department (ED) up to 24 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cutaneous Traction | Skeletal Traction
Number analyzed (Participants) | 37 | 29
minutes | 24 [12 to 50] | 57 [40 to 80]

2. Primary Outcome: Time to Pass Guidewire After Attaining Starting Point
Description: Time to pass guidewire across reduced fracture once opening reamer is used in OR
Time Frame: while in Emergency Department (ED) up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cutaneous Traction | Skeletal Traction
Number analyzed (Participants) | 37 | 29
minutes | 15 (24) | 18 (17)

ADVERSE EVENTS:
Groups:
- Cutaneous Traction: Applied by using a strap on boot that attaches to the leg. A rope is attached to the boot. Weight is attached to the rope to use gravity to pull traction. The traction is left in place until patient is taken to surgery for reduction of the femur fracture.
  Femoral Traction: Temporary intervention to realign the broken bone and help relieve pressure and muscle spasms until operative fixation.
- Skeletal Traction: A small incision is made on the inside of the knee and a pin is surgically inserted through the bone. Weights are then attached that will pull traction on the broken femur. This traction pin will stay in until patient is taken to surgery for reduction of the femur fracture.
  Femoral Traction: Temporary intervention to realign the broken bone and help relieve pressure and muscle spasms until operative fixation.
Arm/Group | Cutaneous Traction | Skeletal Traction
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/29
Other Adverse Events (participants affected / at risk) | 0/37 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cutaneous Traction (N=37) | Skeletal Traction (N=29)
Foot numbness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Foot was numb for 1 day after boot traction applied. Numbness completely resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No